CLINICAL TRIAL: NCT03269071
Title: Neural Stem Cell Transplantation in Multiple Sclerosis Patient: a Phase I Study
Brief Title: Neural Stem Cell Transplantation in Multiple Sclerosis Patients
Acronym: STEMS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Fondazione Italiana Sclerosi Multipla (Other)
Responsible Party: Principal Investigator, Gianvito MARTINO, Prof., IRCCS San Raffaele
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2016-002020-86 (EudraCT)
Record Dates: First submitted 2017-08-30; First posted 2017-08-31 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Progressive Multiple Sclerosis
Keywords: Multiple Sclerosis; Cell Therapy; Human Neural Stem Cells
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment Cohort A (Experimental): See Study Description
  TC-A: 0.7 x 10^6 ± 10% human fetal-derived Neural Stem Cells (hNSCs) / kg of body weight
  Interventions: Drug: human fetal-derived Neural Stem Cells (hNSCs)
- Treatment Cohort B (Experimental): See Study Description
  TC-B: 1.4 x 10^6 ± 10% human fetal-derived Neural Stem Cells (hNSCs) / kg of body weight
  Interventions: Drug: human fetal-derived Neural Stem Cells (hNSCs)
- Treatment Cohort C (Experimental): See Study Description
  TC-C: 2.8 x 10^6 ± 10% human fetal-derived Neural Stem Cells (hNSCs) / kg of body weight
  Interventions: Drug: human fetal-derived Neural Stem Cells (hNSCs)
- Treatment Cohort D (Experimental): See Study Description
  TC-D: 5.7 x 10^6 ± 10% human fetal-derived Neural Stem Cells (hNSCs) / kg of body weight
  Interventions: Drug: human fetal-derived Neural Stem Cells (hNSCs)

INTERVENTIONS:
Drug: human fetal-derived Neural Stem Cells (hNSCs) — The Drug Product (DP) can be classified as an ATIMP belonging to the class of Cell Therapy Medicinal Products (EU law). The ATIMP consists of human fetal-derived Neural Stem Cells (hNSCs) re-suspended in their final formulation medium as defined in the Investigational Medical Product Dossier (IMPD).
  For dosage indications, see specific Treatment Cohorts (TC), from A to D.
  The product will be administered intrathecally through lumbar puncture.
  Other Names: human Neural Stem Cells (hNCSs)

SUMMARY:
This is a phase I study evaluating the feasibility, safety and tolerability of intrathecally administered human Neural Stem Cells (hNSCs), at an escalating dose ranging from 0.7x10^6±10% cells to 5.7x10^6±10% cells/kg of body weight, in patients affected by Progressive Multiple Sclerosis

DETAILED DESCRIPTION:
This is a prospective, monocentric, national, therapeutic exploratory, phase I, not randomized, open label, not controlled, single dose escalation clinical trial.

Each subject will participate in the study for approximately 96 weeks. Participation will include a screening evaluation between -28 and -7 days before the Advance Therapy Investigational Medicinal Products (ATIMP) administration.

A follow-up with clinical visits will be performed from 1 to 96 weeks.

The protocol will consist of a total of four treatment cohorts (TCs), labeled from A to D, each receiving a single escalating dose of allogenic fetal-derived human Neural Stem Cells (hNSCs) injected intrathecally, as it follows:

* TC-A: 0.7x10^6 ± 10% cells/kg of body weight;
* TC-B: 1.4x10^6 ± 10% cells/kg of body weight;
* TC-C: 2.8x10^6 ± 10% cells/kg of body weight;
* TC-D: 5.7x10^6 ± 10% cells/kg of body weight.

The intrathecal injection of hNSCs will be performed in a hospitalized setting. The trial will start with TC-A and will go through the subsequent enrolment of patients to be included in TCs from B to D.

Each cohort will consist of three patients at minimum. In case of safety issue the number in each TC will be increased to six patients.

After the inclusion of the first patient of the TC the investigators will wait at least 14 days to treat the second patient. The same interval time will be used for all the following patient within the same TC. After the inclusion of all the planned patients within a TC and with no Dose Limiting Toxicity (DLT) within the TC, the investigators will wait at least 3 months before switching to the upper TC. In case of 1 DLT within the TC, the cohort will be extended to six patients. If another DLT will be observed, the current dosage will be considered excessive and the immediate lower dosage will be considered the Maximum Tolerated Dose (MTD).

The safety monitoring board will review all safety date in the case of evaluated Adverse Event (AE) ≥ 3 "possibly related to human Neural Stem Cells" by investigators and in any case before the shifts between TCs.

This approach will be repeated for every TC up to the end of the study. At the end of the total follow-up, a long term follow up is planned for all enrolled and treated patients in the study, in accordance with the national applicable laws and the international guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Signature of the informed consent by the patient or patients' legal tutors
2. Age 18 to 55 years
3. Diagnosis of a. Progressive MS as per the revised MC Donald 2010 criteria with a progressive course according to 2013 Lublin phenotypes classification (PMS) with failure or intolerance to all approved therapies according to the disease course or without any alternative approved therapy
4. Evidence of progression of disease defined by an increase of ≥ 0.5 Expanded Disability Status Scale (EDSS) points in the last 12 months
5. Disease duration 2 to 20 years (included)
6. Expanded Disability Status Scale (EDSS) ≥ 6.5
7. Presence of oligoclonal band in the cerebrospinal fluid (CSF) is required for Primary Progressive MS

Exclusion Criteria:

They will be excluded from the study patients:

1. with any active or chronic infection or diseases other than MS including but not limited to infection with HIV1-2, Hepatitis B or Hepatitis C and tuberculosis or immune deficiency syndromes;
2. treated with any immunosuppressive therapy, including but not limited to natalizumab and fingolimod, within the 3 months prior to screening;
3. treated with interferon-beta or glatiramer acetate within the 30 days prior to screening;
4. treated with corticosteroids within the 30 days prior to screening;
5. if relapse occurred during the 30 days prior to screening;
6. with contraindications for or intolerance to any medication, treatments and procedures that will be used in the study;
7. pregnant or in lactation or of childbearing age who are not willing to use a contraceptive method effective* for the entire duration of the study;
8. who, in the opinion of the investigator, showing any condition that would preclude study participation.

   * refer to guideline http://www.hma.eu/fileadmin/dateien/Human_Medicines/01 About_HMA/Working_Groups/CTFG/2014_09_HMA_CTFG_Contraception.pdf

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
SHORT TERM (0-24 hours) Overall survival | 0-24 hours after intrathecal injection of human Neural Stem Cells (hNSCs)
  Number of patients alive all over the trial
SHORT TERM (0-24 hours) Overall safety and tolerability measured by Adverse Event (AE) recording | 0-24 hours after intrathecal injection of human Neural Stem Cells (hNSCs)
  Number of AEs in alive patients all over the trial
SHORT TERM (0-24 hours) Changes in neurological conditions not related to disease | 0-24 hours after intrathecal injection of human Neural Stem Cells (hNSCs)
  Number of changes in neurological conditions not related to disease of alive patients all over the trial
SHORT TERM (0-24 hours) Proportion of successful intrathecal administration procedure (feasibility) | 0-24 hours after intrathecal injection of human Neural Stem Cells (hNSCs)
  Number of successful intrathecal administration procedures versus all intrathecal administration procedures in the whole trial
MID TERM (day 1- day 14) Overall survival | from 1 to 14 days after intrathecal injection of human Neural Stem Cells (hNSCs)
  Number of alive patients in the whole trial
MID TERM (day 1- day 14) Overall safety and tolerability measured by AE recording | from 1 to 14 days after intrathecal injection of human Neural Stem Cells (hNSCs)
  Number of AEs of alive patients in the whole trial
MID TERM (day 1- day 14) Changes in neurological conditions not related to disease | from 1 to 14 days after intrathecal injection of human Neural Stem Cells (hNSCs)
  Number of changes in neurological conditions not related to disease in alive patients of the whole trial
LONG TERM (day 15 - week 96) Overall survival | from day 15 to week 96 after intrathecal injection of human Neural Stem Cells (hNSCs)
  Number of alive patients in the whole trial
LONG TERM (day 15 - week 96) Overall safety and tolerability measured by AE recording | from day 15 to week 96 after intrathecal injection of human Neural Stem Cells (hNSCs)
  Number of AEs in alive patients of the whole trial
Long term incidence of malignancies | from day 0 to week 96 after intrathecal injection of human Neural Stem Cells (hNSCs)
  Incidence of malignancies in alive patients of the whole trial
Evaluation of changes in quality of life measures | 12, 24, 48, 72 and 96 weeks
  Health-related quality of life will be assessed by standardized questionnaires
LONG TERM (day 15 - week 96) Changes in neurological conditions not related to the disease | from day 15 to week 96 after intrathecal injection of human Neural Stem Cells (hNSCs)
  Number of changes in the neurological conditions not related to disease in alive patients of the whole trial

CONTACTS AND LOCATIONS:
Overall Officials: Gianvito Martino, Principal Investigator — IRCCS San Raffaele
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No
It is not yet known the best way to exploit the Individual Participant data (IPD) that will become available

REFERENCES:
- [Result] Kokaia Z, Martino G, Schwartz M, Lindvall O. Cross-talk between neural stem cells and immune cells: the key to better brain repair? Nat Neurosci. 2012 Jul 26;15(8):1078-87. doi: 10.1038/nn.3163. PMID 22837038
- [Result] Martino G, Franklin RJ, Baron Van Evercooren A, Kerr DA; Stem Cells in Multiple Sclerosis (STEMS) Consensus Group. Stem cell transplantation in multiple sclerosis: current status and future prospects. Nat Rev Neurol. 2010 May;6(5):247-55. doi: 10.1038/nrneurol.2010.35. Epub 2010 Apr 20. PMID 20404843
- [Result] Pluchino S, Gritti A, Blezer E, Amadio S, Brambilla E, Borsellino G, Cossetti C, Del Carro U, Comi G, 't Hart B, Vescovi A, Martino G. Human neural stem cells ameliorate autoimmune encephalomyelitis in non-human primates. Ann Neurol. 2009 Sep;66(3):343-54. doi: 10.1002/ana.21745. PMID 19798728
- [Result] Pluchino S, Quattrini A, Brambilla E, Gritti A, Salani G, Dina G, Galli R, Del Carro U, Amadio S, Bergami A, Furlan R, Comi G, Vescovi AL, Martino G. Injection of adult neurospheres induces recovery in a chronic model of multiple sclerosis. Nature. 2003 Apr 17;422(6933):688-94. doi: 10.1038/nature01552. PMID 12700753
- [Result] Pluchino S, Zanotti L, Rossi B, Brambilla E, Ottoboni L, Salani G, Martinello M, Cattalini A, Bergami A, Furlan R, Comi G, Constantin G, Martino G. Neurosphere-derived multipotent precursors promote neuroprotection by an immunomodulatory mechanism. Nature. 2005 Jul 14;436(7048):266-71. doi: 10.1038/nature03889. PMID 16015332
- [Derived] Genchi A, Brambilla E, Sangalli F, Radaelli M, Bacigaluppi M, Furlan R, Andolfo A, Drago D, Magagnotti C, Scotti GM, Greco R, Vezzulli P, Ottoboni L, Bonopane M, Capilupo D, Ruffini F, Belotti D, Cabiati B, Cesana S, Matera G, Leocani L, Martinelli V, Moiola L, Vago L, Panina-Bordignon P, Falini A, Ciceri F, Uglietti A, Sormani MP, Comi G, Battaglia MA, Rocca MA, Storelli L, Pagani E, Gaipa G, Martino G. Neural stem cell transplantation in patients with progressive multiple sclerosis: an open-label, phase 1 study. Nat Med. 2023 Jan;29(1):75-85. doi: 10.1038/s41591-022-02097-3. Epub 2023 Jan 9. PMID 36624312

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-10): https://cdn.clinicaltrials.gov/large-docs/71/NCT03269071/Prot_SAP_000.pdf